CLINICAL TRIAL: NCT03082677
Title: Open Label Phase II Study of Ixazomib for the Prevention of Recurrent or Late Acute and Chronic Graft-versus-Host Disease at 1-year After Allogeneic Hematopoietic Stem Cell Transplantation in Patients With Hematologic Malignancies
Brief Title: Study of Ixazomib to Prevent Recurrent or Late Acute and Chronic Graft-versus-Host Disease 1-year After Allogeneic Hematopoietic Stem Cell Transplantation in Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Millennium: The Takeda Oncology Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-076
Record Dates: First submitted 2017-03-13; First posted 2017-03-17 (Actual); Results first posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2021-09

CONDITIONS: Myeloid Hematologic Malignancy; Lymphoid Hematologic Malignancy
Keywords: Ixazomib; Graft-versus-Host Disease; Allogeneic Hematopoietic Stem Cell Transplantation; 16-076
MeSH Terms: conditions — Graft vs Host Disease | interventions — ixazomib

STUDY DESIGN:
Intervention Model Description: This is a single arm phase 2 study to evaluate a post-transplant proteasome inhibitor, ixazomib, as prophylaxis against recurrent or late acute and chronic GVHD. Ixazomib will be initiated within days 100 to 150 post-transplant in patient's ≥ 18 years-old with either myeloid or lymphoid hematologic malignancy treated with a RI or NMA HSCT and will have received calcineurin inhibitor based drug (tacrolimus or cyclosporin) and methotrexate as part of their initial GVHD prophylaxis.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ixazomib (Experimental): Ixazomib beginning between day +100 to +150 at a dose of 4 mg orally once per week (3 weeks on/ 1 week off). The patients will continue on this same dose until taper off from immunosuppressants or 1 year post-HSCT is reached (whichever occurs first) or until the patient develops GVHD or malignant disease relapse/progression occurs.
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Ixazomib — Ixazomib beginning between day +100 to +150 at a dose of 4 mg orally once per week (3 weeks on/ 1 week off).
  Other Names: MLN 9708

SUMMARY:
This is a single arm open label phase 2 study evaluating the potential effect of ixazomib on the prevention of recurrent or late acute graft-versus-host disease (GVHD) and chronic GVHD at 1-year following reduced intensity (RI) or non-myeloablative (NMA) allogeneic hematopoietic stem cell transplantation (HSCT) for the treatment of hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older.
* Diagnosis: myeloid or lymphoid hematologic malignancy treated with a RI or NMA conditioning HSCT who received calcineurin inhibitor based drug (for example: tacrolimus or cyclosporin) and methotrexate as part of their initial GVHD prophylaxis. Patients who received sirolimus as part of their GVHD prophylaxis will be eligible.
* Recipients of 8-7/8 HLA-matched donor. Post-HSCT period within day +100 to day +150.
* Female patients who:

  * Are postmenopausal for at least 1 year before the screening visit, OR
  * Are surgically sterile, OR
  * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence and withdrawal are not acceptable methods of contraception).
* Male patients, even if surgically sterilized (i.e. Status post-vasectomy) must agree to one of the following:

  * Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject (periodic abstinence and withdrawal are not acceptable methods of contraception).
* Organ Function and Performance Status Criteria:
* Karnofsky score ≥ 70 %
* Absolute neutrophil count (ANC) ≥ 1000/mm3 and platelet count ≥ 75,000/mm3. Platelet transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.
* Calculated creatinine clearance ≥ 30 mL/min (based on the Cockcroft and Gault method)
* Total bilirubin ≤ 1.5 x upper limit of normal range (ULN).
* AST/ALT ≤ 3 x ULN (unless benign congenital hyperbilirubinemia).
* Hemoglobin > 8.0 g/dL. Red blood cell transfusions to help patients meet eligibility criteria are not allowed within 3 days before study enrollment.

Exclusion Criteria:

* Disease: evidence of progressive disease at the time of study enrollment.
* Prior Therapy: one or more prior allogeneic stem cell transplantation (prior autologous transplant is acceptable).
* Active acute or chronic GVHD.
* Active and uncontrolled infection.
* Pregnant or breast feeding.
* Major surgery within 14 days before enrollment.
* Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
* Systemic treatment, within 14 days before the first dose of ixazomib, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Patient or guardian unable to give informed consent or unable to comply with the treatment protocol including appropriate supportive care, follow-up and research tests.
* Patients with known allergy to boron or boron-containing products, or excipients in the various formulations of any agent.
* Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Patient with ≥ Grade 3 peripheral neuropathy, or Grade 2 with pain on clinical examination during the screening period.
* Received post-transplant cyclophosphamide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2021-09-02 (Actual); Study Completion 2021-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doris M Ponce, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ixazomib
Started | 20
Completed | 18
Not Completed | 2
Not completed — Not Treated | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ixazomib
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 59 [45 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Absence of Grade II-IV aGVHD or Chronic GVHD Diagnostic Features
Description: Therapeutic response will be determined by the absence of grade II-IV aGVHD or chronic GVHD diagnostic features.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Ixazomib
Number analyzed (Participants) | 18
Participants
  No aGCHD or cGVHD | 13
  aGCHD or cGVHD | 5

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Ixazomib
All-Cause Mortality (participants affected / at risk) | 2/18
Serious Adverse Events (participants affected / at risk) | 2/18
Other Adverse Events (participants affected / at risk) | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib (N=18)
Fever (General disorders) | 1
Lung infection (Infections and infestations) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Vasovagal reaction (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixazomib (N=18)
Anemia (Blood and lymphatic system disorders) | 9
APTT time prolonged (Investigations) | 1
Lymphopenia (Blood and lymphatic system disorders) | 6
Neutropenia (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 9
Chest pain (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Peripheral edema (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Mouth pain (Gastrointestinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 1
Post-nasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Conjunctivitis (Infections and infestations) | 1
Eye pain (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Elevated alanine aminotransferase (Investigations) | 8
Elevated alkaline phosphatase (Investigations) | 1
Elevated aspartate aminotransferase (Investigations) | 11
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 8
Dysgeusia (Nervous system disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
GERD (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Pain (General disorders) | 2
Weight Gain (General disorders) | 1
Bronchial infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Skin infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Cholesterol high (Investigations) | 5
Creatinine increased (Investigations) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 13
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 6
Hypernatremia (Metabolism and nutrition disorders) | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 2
Vaginal discharge (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Xerodermia (Skin and subcutaneous tissue disorders) | 2
Pruritis (Skin and subcutaneous tissue disorders) | 1
Rash, acneiform (Skin and subcutaneous tissue disorders) | 2
Rash, maculo-papular (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-09): https://cdn.clinicaltrials.gov/large-docs/77/NCT03082677/Prot_SAP_000.pdf